CLINICAL TRIAL: NCT04436302
Title: The Efficacy of Exergaming in People With Major Neurocognitive Disorder Residing in Long-term Care Facilities: A Randomized Controlled Trial
Brief Title: Exergaming in People With Major Neurocognitive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Davy Vancampfort (Other)
Responsible Party: Sponsor-Investigator, Davy Vancampfort, Professor, KU Leuven
Organization: KU Leuven (Other)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 042020
Record Dates: First submitted 2020-06-03; First posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Randomised Controlled Trial; Major Neurocognitive Disorder; Long-term Care Facility; Physical Activity; Cognitive Impairment
MeSH Terms: conditions — Motor Activity; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Dividat senso exergame device
  Interventions: Device: Exergame device
- Control (Active Comparator): Listening to music
  Interventions: Device: Exergame device

INTERVENTIONS:
Device: Exergame device — motor-cognitive training
  Other Names: Dividat senso

SUMMARY:
This randomized controlled trial explores the efficacy of an 8-week standing exergaming program in people with major neurocognitive disorder (MNCD) residing in long-term care facilities.

DETAILED DESCRIPTION:
This randomized controlled trial explores the efficacy of an 8-week standing exergaming program in people with major neurocognitive disorder (MNCD) residing in long-term care facilities. Fifty inpatients with mild to moderate MNCD will be randomly assigned to three times weekly for eight weeks 15 min of exergaming versus watching preferred music videos. The Montréal Cognitive Assessment (MoCA), Short Physical Performance Battery (SPPB), Neuropsychiatric Inventory (NPI), Cornell Scale for Depression in Dementia (CSDD), Dementia Quality of Life (DQoL), Katz activities of daily living (ADL) and Instrumental ADL (IADL) are measured at baseline and post intervention.

ELIGIBILITY:
Inclusion criteria included:

* a Diagnostic and Statistical Manual of Mental Disorders (DSM) 5 diagnosis of MNCD (American Psychiatric Association, 2013)
* aged 65 years or older
* a score of minimum 10 on the Mini-Mental State Examination (MMSE)
* residing at least two weeks in the care facility at the time of inclusion
* being physically capable of doing standing exercises (whether or not with extra support).

Possible causes of MNCD were vascular dementia, Alzheimer's disease, mixed dementia, Parkinson's disease or Lewy body disease.

Exclusion criteria consisted of:

* any unstable cardiovascular or other health condition which according to the American College of Sports Medicine Standards might lead to unsafe participation
* a score lower than 10 on the MMSE
* a planned transfer to another setting within the following two months.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-01-02 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
MoCA | 2 years
  Montréal Cognitive Assessment
SPPB | 2 years
  Short Physical Performance Battery
NPI | 2 years
  Neuropsychiatric Inventory
CSDD | 2 years
  Cornell Scale for Depression in Dementia
DQOL | 2 years
  Dementia Quality of Life
(I)ADL | 2 years
  Activities of daily living

CONTACTS AND LOCATIONS:
Locations (1):
- Long-term care facility 'de Wingerd', Leuven, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Swinnen N, Vandenbulcke M, de Bruin ED, Akkerman R, Stubbs B, Firth J, Vancampfort D. The efficacy of exergaming in people with major neurocognitive disorder residing in long-term care facilities: a pilot randomized controlled trial. Alzheimers Res Ther. 2021 Mar 30;13(1):70. doi: 10.1186/s13195-021-00806-7. PMID 33785077